CLINICAL TRIAL: NCT07373483
Title: Interactive Electronic Devices (IEDs) in the Home: Exploring How Young Children Use IEDs in the Family Home Setting
Brief Title: Observing 3-5 Year Old Children's Use of Interactive Electronic Devices (IED) in the Family Home to Understand the Context These Devices Are Being Used in, Exploring Whether Socioeconomic Factors or Parent's Own Use of Such Devices Influence the Child's IED Usage.
Acronym: iKids
Status: Recruiting | Type: Observational
Sponsor: Sheffield Hallam University (Other)
Collaborators: University of Chester (Other)
Responsible Party: Sponsor
Other Study IDs: AA63081485; NIHR159040 (Other Grant/Funding Number: NIHR - National Institute for Health and Care Research)
Record Dates: First submitted 2025-12-05; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: This Study Explores How Young Children Aged 3 to 5 Use Interactive Electronic Devices
Keywords: Early Years; Mobile Devices; Socioeconomic Development; Home Context

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Population: Children aged 3-5 years old: We will be recruiting participants who are 3-5 years of age and use interactive electronic devices and who have not been clinically diagnosed with a developmental disorder by a medical professional.
- Study Population: Parent of children aged 3-5 years involved in the study: We will interview a parent or carer of the 3-5 year old children involved in the study to gain insights from the video recordings taken of their children using interactive electronic devices in the family home.

SUMMARY:
This study aims to explore the context of how children aged 3-5 use interactive electronic devices like tablets or smartphones in their everyday home environment. The researchers will look at the social, family, and environmental factors that shape this use.

This study will use a qualitative ethnographic approach to explore how young children aged 3-5 use interactive electronic devices (IEDs) in the home. Data will be collected through questionnaires, exploring parent and child IED use, and video recordings of children in their natural home environment over one week, with three recording sessions of approximately four hours each. Following the recording period, selected clips will be reviewed with parents during a semi-structured interview to reflect on behaviours, routines, and context.

These videos will help capture not just what children do, but also how they interact with others while using the devices - like gestures, facial expressions, and conversations. The researchers will process the data and extract some video clips. These clips will be used to discuss with parents what they saw in the videos during 60-90-minute interviews to get their insights and giving us a deeper understanding of the child's behaviour and communication.

Data analysis will involve inductive thematic analysis of interview transcripts to identify patterns and themes in parental reflections and experiences. To support and accelerate this process, video analysis will be used to extract key moments and behaviours from the recordings, helping to contextualise and enrich the thematic findings. This combined approach will allow for a deep understanding of the social and environmental factors shaping children's technology use.

The study will include families from a range of socioeconomic backgrounds, with children aged 3-5 years of age. Participants will be recruited through early years settings, as well as via flyers distributed across family hubs, community centres, libraries and on social media throughout Yorkshire.

DETAILED DESCRIPTION:
Background:

Interactive electronic devices (IEDs), which the researchers define as any portable screen, such as tablets or mobile phones, are ubiquitous in young children's lives, with 90% of children aged 3-4 years going online. National and international guidelines report a lack of understanding around the family circumstances of when young children are using such devices, limiting recommendations. Few studies have focused on how and when young children use IEDs, and fewer still explore the socioeconomic relationship and IED use of children (Arabiat et al., 2023; Radesky et al., 2020). In conversations with early years practitioners, parents and policymakers, they recognise IEDs as a valuable resource for early years learning, observing how most families from all backgrounds now allow their children to use IEDs (Azevedo et al., 2025). However, what is unknown is how children and their parents are using IEDs and whether there is an observable difference or indeed what circumstances increase or reduce IED usage.

Few studies have examined the experience of young children engaging in screen-based activities.

Studies found that parents advise children to use devices for multiple purposes, such as education and distraction, particularly when parents need to do household chores (Bentley et al., 2016). Studies have also reported contrasting views on the need to establish rules, while many agreed that mobile devices are an unavoidable part of modern life (Kabali et al., 2015).

However, to date, the researchers are unaware of any study that has observed children in their home environment to better understand their behaviours and interactions with mobile devices.

Research Aim:

This study aims to explore how young children (aged 3-5) use interactive electronic devices like tablets or smartphones in their everyday home environment. The researchers will look at the social, family, and environmental factors that shape this use.

Main research question: What is the context and nature of interactions in which children use IEDs in their home environment?

1. How do young children aged 3-5 use interactive electronic devices within the routines and relationships of their family home?
2. In what ways do family structure, financial circumstances, and cultural background influence the nature and context of children's IED use?
3. How do parents perceive the role of IED in supporting or challenging their caregiving practices, including supervision, learning, and daily household management?

Methods:

This ethnographic study will adopt a qualitative and pragmatic approach (Morgan, 2014), to explore the social, familial and environmental contexts in which young children use interactive electronic devices (IEDs) at home.

The researchers will employ video-reflexive ethnography (VRE), which combines video ethnography - capturing routine behaviours and interactions of children using IEDs in the home - with video-reflexivity, involving interviews with parents to reflect on these behaviours (Korstjens et al., 2021). Video recordings will provide rich data on children's practices and behaviours related to IED use (Manojlovich et al., 2019), offering access to verbal and non-verbal communication (Risley and Hart, 1968) and insights into the interplay of multiple communication channels (Heath et al., 2007). Engaging parents/carers in interpreting these observations will enhance the visibility of these interactions and allow reflection on the child's lived experiences (Gordon et al., 2017).

Participants and Recruitment:

Eligible families must have a child aged 3-5 years with no diagnosed developmental disorders. The study will be promoted using posters placed in family-oriented locations such as libraries, community centres, family hubs, and leisure centres. To ensure socioeconomic diversity, nurseries, family hubs, and community centres will be selected from areas in both the highest and lowest IMD quintiles in the West Yorkshire region. The researchers aim to recruit 20 parents/carers - 10 from low-income areas and 10 from high-income areas.

Families will be provided with contact details for the lead researcher and reassured that they may withdraw from the study at any time. This process prioritises openness, trust, and informed consent.

As this study is part of a wider NIHR -funded research project, the researchers will use the contacts established with different stakeholders (Local Authorities, Early Years Settings) and participants to advertise and recruit participants.

Parents/carers of children aged 3-5 are directed to a weblink where they can read more about the study and express interest to meet the researcher and learn more about the study. Parents/carers will be offered to meet ahead of agreeing to partake in the research and given the opportunity to ask any questions they have, learn more about the research project, and meet the researcher who will be coming into their home to place the cameras and interview them.

A recent systematic review (Hennink & Kaiser, 2022) suggests that 9-17 interviews are sufficient for relatively homogeneous populations, although some argue that sample size should be determined during analysis. Taking a pragmatic approach, the researchers believe this sample size will allow us to reach thematic saturation.

To better understand participant demographics, the researchers will collect data on age, gender, ethnicity, marital status, parenthood, and years of education as well as additional demographic information - such as family structure, cultural background, and financial and educational context. The questionnaire will also ask about the child's and parent's own use of interactive electronic devices by using the screen Q and SAS-SV questionnaires. A combined version of these questionnaires will be sent to parents before the camera is placed in their home. The answers to the questionnaire will guide the interview questions and prompt conversation around the observations from the video and sound recordings.

Data Collection, Processing, and Analysis:

Video recording within the home environment presents several challenges, including its resource-intensive nature, potential influence on participant behaviour (Asan and Montague, 2014), and concerns around privacy (Everri et al., 2020). To address these issues thoughtfully and ethically, the researchers will begin with family engagement meetings, where they will discuss key topics such as participant rights, data anonymisation, privacy protection, and the intended use of recorded material.

Recognising the sensitive nature of placing a camera in the family home, the researchers will also offer families the opportunity for individual follow-up meetings after the group engagement sessions. These one-to-one conversations - held in a location of the participant's choosing, such as a local café or community space - are intended to foster trust and build rapport between researchers and families. By creating a more informal and personalised setting, the researchers hope to support open dialogue and ensure families feel comfortable and confident in their participation.

A video camera will be placed in a communal room (e.g., a sitting room) within the family home for a period of seven days. However, to minimise self-consciousness and reduce the impact of observation on behaviour, recording will only take place during the final three days - ideally, over two weekdays and one weekend day. Parents and carers will be actively involved in determining the most appropriate location for the camera, ensuring it is placed in a space where the child spends time and feels comfortable.

To maintain flexibility and reduce intrusiveness, the family will have the ability to turn the camera on and off or cover the camera lens. If any footage is captured that parents feel is inappropriate or outside the scope of the study, they may request its removal. To facilitate this, families will be provided with a diary and a deletion request form. These tools will allow parents to note specific times and dates they wish to exclude from the final dataset - for example, if the camera was left on after the child stopped using the IED. Alternatively, requests can be submitted during the data processing stage, and the relevant clips will be removed without being viewed.

During data processing, a member of the research team will review all footage and automatically delete any segments where the child is not present. This approach ensures that only relevant interactions are retained and respects the privacy and autonomy of participating families.

Interview transcripts and video data will be anonymised during analysis, with names and other identifying details removed or replaced with pseudonyms. Only the research team at Sheffield Hallam University will have access to identifiable data.

All data will be stored securely on encrypted devices and institutional servers, in accordance with the Data Protection Act (2018). Anonymised data will be archived in the Sheffield Hallam Research Data Archive for up to 10 years following the last third-party access request. Paper documents will be stored in locked cabinets and securely disposed of at the end of the retention period. Participants may withdraw at any time, and their data can be removed up until June 2026.

From the recordings, the researchers will select up to ten 3-minute clips featuring the child interacting with IEDs and family or friends. The PI and RF will review these clips, asking "What is 'this' an example of?" and use open coding to develop themes (Khandkar, 2009). A subsample size of 20% of the video footage will be reviewed by two other members of the research team, offering opportunity for agreement on what the researchers are looking before moving on to the full sample. Rather than simply describing events, researchers will interpret the meaning behind them (Goldman, 2014).

These clips will be shown to parents/carers during reflective semi-structured interviews, allowing them to share their interpretations. Interviews will follow a guide with open-ended questions, informed by the completed questionnaire, using reflective listening. To promote reflexivity, the researchers will pause the video at key moments and ask interview questions.

Each interview will last approximately 60-90 minutes, be digitally recorded with consent, and transcribed verbatim. Identifiable information will be removed, and pseudonyms assigned to ensure confidentiality. Transcripts will be imported into Nvivo 12 for analysis.

The researchers will use inductive thematic analysis to interpret the data (Clarke et al., 2015), acknowledging that researchers' prior knowledge may influence theme development (Maggs-Rapport, 2000). To mitigate this, four members of the research team will review at least 20% of the same videos before coming to an agreement of what to measure and the PI and RF will then independently conduct the analysis over the rest of the videoclips and then will convene to discuss emerging themes. The researchers will include extensive participant quotations to support transparency and allow readers to interpret the findings (Eldh et al., 2020).

Data from both the video ethnography and the video-reflexivity interviews will be integrated to provide a rich, contextual understanding of how young children engage with interactive electronic devices (IEDs) and how parents/carers interpret and respond to this use. The video ethnography will offer direct observational insights into children's behaviours, interactions, and environments, while the reflexive interviews will add depth by capturing parental perspectives, contextual explanations, and emotional responses to the footage.

To ensure transparency and rigour in reporting, the researchers will explicitly describe how these two data sources are merged during the analysis phase. This will include outlining the process of cross-referencing coded video segments with interview transcripts, identifying converging and diverging themes, and explaining how parental interpretations either reinforce or challenge the observational data. This triangulation will strengthen the validity of our findings and allow us to explore the interplay between observed behaviour and parental meaning-making (Skivington et al., 2021).

In the researchers final reporting, they will include a dedicated section detailing the data integration strategy, including examples of how specific video observations were interpreted and expanded upon through parental interviews. This will help readers understand the analytical process and the rationale behind theme development, ensuring clarity and coherence in how the findings are presented.

ELIGIBILITY:
Inclusion Criteria:

* Children between 3 and 5 years old
* Children who use an interactive electronic device
* Children who have received parent/carer consent for participation and provided verbal assent

Exclusion Criteria:

* Children whose parents do not speak and/or understand English
* Children who have been clinically diagnosed with a developmental disorder by a medical professional prior to either baseline or follow-up assessments

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 3-5 year old children, living in Yorkshire, UK, who currently uses an interactive electronic device while at home, without a diagnosed behavioural or cognitive condition.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Ethnographic Observation of Children's use of Interactive Electronic Devices | Through study completion, an average of 6 months.
  Parents' perceptions and attitudes toward their child's use of interactive electronic devices (IEDs) will be assessed through semi-structured interviews. These interviews will explore parents' views on the appropriateness, benefits, and potential risks of IED usage, as well as their beliefs about the circumstances under which their child engages with these devices. Responses will provide qualitative insights into parental attitudes and perceived influences on Early Years children's technology use.
Video Observation | During analysis of video footage (first 3 weeks of participation).
  Video observations made by the researchers will help to provide understanding on how and why the phenomena (child's use of interactive electronic device) occur. Three four hour clips will be selected to analyse for themes and repeated behaviours during the child's device use.

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Craig, PhD, Principal Investigator — Sheffield Hallam University; Liane Beretta de Azevedo, Study Chair — Sheffield Hallam University
Locations (1):
- Sheffield Hallam University, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared via a repository, and requests can be made directly to the Sheffield Hallam Research Data Archive (SHURDA), email address: library-research-support@shu.ac.uk.
  If data is requested during the project period, a data-sharing agreement will be issued between Sheffield Hallam University and the data requester. In this case, data sharing will be restricted to ensure it does not impact the research team's publication plan.
  Fully anonymised data will be stored in SHURDA and be retained for 10 years from the last time a third party requested access.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Hennink, M. and Kaiser, B.N., 2022. Sample sizes for saturation in qualitative research: A systematic review of empirical tests. Social science & medicine, 292, p.114523.
- [Background] Azevedo, L.B., Downes, M., Eastburn, S., Covell, J. and Bissell, P. (2025) 'Early years practitioners' and public health consultants' perspectives on the use of interactive electronic devices in young children: A qualitative study', Child Care Health and Development, 51(1), e70022. doi:10.1111/cch.70022.
- [Background] Bentley, G.F., Turner, K.M. and Jago, R. (2016) 'Mothers' views of their preschool child's screen-viewing behaviour: a qualitative study', BMC Public Health, 16, Article 718. doi:10.1186/s12889-016-3440-z.
- [Background] Clarke, V., Braun, V. and Hayfield, N. (2015) 'Thematic analysis', in Smith, J.A. (ed.) Qualitative Psychology: A Practical Guide to Research Methods. 3rd edn. London: Sage, pp. 222-248.
- [Background] Eldh, A.C., Årestedt, L. and Berterö, C. (2020) 'Quotations in qualitative studies: reflections on constituents, custom, and purpose', International Journal of Qualitative Methods, 19, pp. 1-8. doi:10.1177/1609406920969268.
- [Background] Everri, M., Heitmayer, M., Yamin-Slotkus, P. and Lahlou, S. (2020) 'Ethical challenges of using video for qualitative research and ethnography', in Challenges and Solutions in Ethnographic Research. Abingdon: Routledge, pp. 68-83.
- [Background] Goldman, R. (2014) 'Video representations and the perspectivity framework: Epistemology, ethnography, evaluation, and ethics', in Goldman, R., Pea, R., Barron, B. and Derry, S. (eds.) Video Research in the Learning Sciences. Abingdon: Routledge, pp. 3-37.
- [Background] Heath, C., Luff, P. and Svensson, M.S. (2007) 'Video and qualitative research: analysing medical practice and interaction', Medical Education, 41(1), pp. 109-116. doi:10.1111/j.1365-2929.2006.02641.x.
- [Background] Kabali, H.K., Irigoyen, M.M., Nunez-Davis, R., Budacki, J.G., Mohanty, S.H., Leister, K.P. and Bonner, R.L. Jr. (2015) 'Exposure and use of mobile media devices by young children', Pediatrics, 136(6), pp. 1044-1050. doi:10.1542/peds.2015-2151.
- [Background] Khandkar, S.H. (2009) Open coding. University of Calgary. Available at: https://studylib.net/doc/18074044/open-coding---university-of-calgary (Accessed: 25.11.25).
- [Background] Korstjens, I., Mesman, J., van Helmond, I., de Vries, R. and Nieuwenhuijze, M. (2021) 'The paradoxes of communication and collaboration in maternity care: A video-reflexivity study with professionals and parents', Women and Birth, 34(2), pp. 145-153. doi:10.1016/j.wombi.2020.01.014.
- [Background] Maggs-Rapport, F. (2000) 'Combining methodological approaches in research: ethnography and interpretive phenomenology', Journal of Advanced Nursing, 31(1), pp. 219-225. doi:10.1046/j.1365-2648.2000.01243.x.
- [Background] Manojlovich, M., Frankel, R.M., Harrod, M., Heshmati, A., Hofer, T., Umberfield, E. et al. (2019) 'Formative evaluation of the video reflexive ethnography method, as applied to the physician-nurse dyad', BMJ Quality & Safety, 28(2), pp. 160-166. doi:10.1136/bmjqs-2018-008390.
- [Background] Skivington, K., Matthews, L., Simpson, S.A., Craig, P., Baird, J., Blazeby, J.M. et al. (2021) 'A new framework for developing and evaluating complex interventions: update of Medical Research Council guidance', BMJ, 374, n2061. doi:10.1136/bmj.n2061.
- [Background] Risley, T.R. and Hart, B. (1968) 'Developing correspondence between the non-verbal and verbal behavior of preschool children', Journal of Applied Behavior Analysis, 1(4), pp. 267-281. doi:10.1901/jaba.1968.1-267.
- [Background] Radesky, J.S., Weeks, H.M., Ball, R., Schaller, A., Yeo, S., Durnez, J. et al. (2020) 'Young children's use of smartphones and tablets', Pediatrics, 146(1), e20193518. doi:10.1542/peds.2019-3518.
- [Background] Morgan, D.L. (2014) 'Pragmatism as a paradigm for social research', Qualitative Inquiry, 20(8), pp. 1045-1053. doi:10.1177/1077800413513733.
- [Background] Asan, O. and Montague, E. (2014) 'Using video-based observation research methods in primary care health encounters to evaluate complex interactions', Informatics in Primary Care, 21(4), pp. 161-170. doi:10.14236/jhi.v21i4.72.
- [Background] Arabiat, D., Al Jabery, M., Robinson, S., Whitehead, L. and Mörelius, E. (2023) 'Interactive technology use and child development: A systematic review', Child Care Health and Development, 49(4), pp. 679-715. doi:10.1111/cch.13082.